CLINICAL TRIAL: NCT05548842
Title: Evaluation of Efficacy and Safety of the Combined Seed Extracts of Cassia Obtusifolia Linne and Foeniculum Vulgare Mill in Patients With Chronic Constipation: a Double-blind, Randomized, Placebo-controlled Study
Brief Title: The Combined Seed Extracts of Cassia Obtusifolia Linne and Foeniculum Vulgare Mill in Patients With Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2022-010
Record Dates: First submitted 2022-09-14; First posted 2022-09-22 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Chronic Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined group (Experimental): This group takes the combined seed extracts of Cassia obtusifolia Linne and Foeniculum vulgare Mill for 12 weeks.
  Interventions: Dietary Supplement: The combined seed extracts of Cassia obtusifolia Linne and Foeniculum vulgare Mill
- Placebo group (Placebo Comparator): This group takes placebo for 12 weeks.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: The combined seed extracts of Cassia obtusifolia Linne and Foeniculum vulgare Mill — The combined seed extracts of Cassia obtusifolia Linne and Foeniculum vulgare Mill 1,000 mg/day for 4 weeks
  Arms: Combined group
Dietary Supplement: Placebo group — Placebo 1,000 mg/day for 4 weeks
  Arms: Placebo group

SUMMARY:
The investigators will conduct a randomized, double-blind, placebo-controlled study to investigate the effects and safety of the combination seed extracts of Cassia obtusifolia Linne and Foeniculum vulgare Mill in patients with chronic constipation for 4 weeks.

DETAILED DESCRIPTION:
A previous animal study has indicated that the combined seed extracts of Cassia obtusifolia Linne and Foeniculum vulgare Mill have a laxative effect by recovering stool parameters, colonic morphology, and activation of mAchRs and their downstream signaling pathway in constipation. Furthermore, this study provides that the combined seed extracts of Cassia obtusifolia Linne and Foeniculum vulgare Mill could be considered as a therapeutic drug candidate for the prevention or treatment of constipation. Therefore, the investigators a randomized, double-blind, placebo-controlled study to investigate the effects and safety of the combination seed extracts of Cassia obtusifolia Linne and Foeniculum vulgare Mill in patients with chronic constipation for 4 weeks. The Investigators examine stool transit time, constipation Visual Analogue Scale (VAS), Bristol stool Form scale type 3 and 4 (frequency per week), VAS for Irritable Bowel Syndrome (VAS-IBS) questionnaire, IBS severity scoring system, BS Quality of Life instrument at baseline, as well as after 2 and 4 weeks of intervention. Interferon-1β and tumor necrosis factor-α concentrations were measured at baseline and 4 weeks. One hundred adults were administered either 1,000 mg of the combined seed extracts of Cassia obtusifolia Linne and Foeniculum vulgare Mill or a placebo each day for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

*Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis

**Must include two or more of the following:

* Straining during more than ¼ (25%) of defecations
* Lumpy or hard stools (Bristol Stool Form Scale 1-2) more than ¼ (25%) of defecations
* Sensation of incomplete evacuation more than ¼ (25%) of defecations
* Sensation of anorectal obstruction/blockage more than ¼ (25%) of defecations
* Manual maneuvers to facilitate more than ¼ (25%) of defecations (e.g., digital evacuation, support of the pelvic floor)
* Fewer than three spontaneous bowel movements per week
* Loose stools are rarely present without the use of laxatives
* Insufficient criteria for irritable bowel syndrome

Exclusion Criteria:

* A person who is taking a constipation treatment prescribed by a doctor within 1 month from the date of screening
* Those who have been taking lactobacillus or probiotics within the last 1 month
* Those with secondary constipation induced by drugs or diseases.
* Abnormal liver or renal function (more than twice the normal upper limit of the research institute)
* Uncontrolled diabetes mellitus (>160 mg/dL of fasting blood sugar)
* Uncontrolled hypertension (>160/100 mmHg)
* Uncontrolled thyroid diseases.
* Those who are taking drugs, functional foods, herbs, etc. that may affect depression
* Alcohol abuser
* Allergic reaction to this test food
* Those who participated in other drug clinical trials within 1 month from the screening date.
* Severe gastrointestinal symptoms such as heartburn and indigestion
* Those who are pregnant, lactating, or plan to become pregnant during the clinical trial
* Those who are judged to be unsuitable by the PI for other reasons

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Colonic transit time during 2 weeks | At the 2nd weeks after the start of the study
  The number of retained radiopaque markers on a Day 4 plain abdominal film
Change in Colonic transit time during 4 weeks | At the 4th weeks after the start of the study
  The number of retained radiopaque markers on a Day 4 plain abdominal film

SECONDARY OUTCOMES:
Change in Constipation Visual Analogue Scale during 2 weeks | At the 2nd weeks after the start of the study
  The minimum score was 0, the maximum score was 100, and higher scores mean a worse outcome.
Change in Bristol stool Form scale type 3 and 4 (frequency per week) during 2 weeks | At the 2nd weeks after the start of the study
  Frequency of Bristol stool Form scale types 3 and 4 per week
Change in Visual Analogue Scale for Irritable Bowel Syndrome during 2 weeks | At the 2nd weeks after the start of the study
  All except item 1 are rated from 0 to 100 points using the Visual Analogue Scale. A total of 700 points is obtained. Higher scores mean a better outcome.
Change in Irritable Bowel Syndrome severity scoring system during 2 weeks | At the 2nd weeks after the start of the study
  Among the questions, categorical questions asking about abdominal pain or bloating are excluded from the score calculation, and the remaining 5 questions are rated from 0 to 100 points using the Visual Analogue Scale. The total score is 500 points. Higher scores mean a worse outcome.
Change in Irritable Bowel Syndrome Quality of Life instrument during 2 weeks | At the 2nd weeks after the start of the study
  5 points for 'not at all', 4 points for 'somewhat', 3 points for 'moderate', 2 points for 'very much', and 1 point for 'severe' (i.e., count opposite the number on the questionnaire). Higher scores indicate higher quality of life.
Change in Interferon-1β during 4 weeks | At 4th weeks after the start of the study
  concentration (U/ml)
Change in Tumor necrosis factor-α during 4 weeks | At 4th weeks after the start of the study
  concentration (pg/ml)
Change in Constipation Visual Analogue Scale during 4 weeks | At the 4th weeks after the start of the study
  The minimum score was 0, the maximum score was 100, and higher scores
Change in Bristol stool Form scale type 3 and 4 (frequency per week) during 4 weeks | At the 4th weeks after the start of the study
  Frequency of Bristol stool Form scale types 3 and 4 per week
Change in Visual Analogue Scale for Irritable Bowel Syndrome during 4 weeks | At the 4th weeks after the start of the study
  All except item 1 are rated from 0 to 100 points using the Visual Analogue Scale. A total of 700 points is obtained. Higher scores mean a better outcome.
Change in Irritable Bowel Syndrome severity scoring system during 4 weeks | At the 4th weeks after the start of the study
  Among the questions, categorical questions asking about abdominal pain or bloating are excluded from the score calculation, and the remaining 5 questions are rated from 0 to 100 points using the Visual Analogue Scale. The total score is 500 points. Higher scores mean a worse outcome.
Change in Irritable Bowel Syndrome Quality of Life instrument during 4 weeks | At the 4th weeks after the start of the study
  5 points for 'not at all', 4 points for 'somewhat', 3 points for 'moderate', 2 points for 'very much', and 1 point for 'severe' (i.e., count opposite the number on the questionnaire). Higher scores indicate higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea